CLINICAL TRIAL: NCT00632515
Title: Screening and Risk Communication for First Degree Relatives of Colorectal Cancer Patients
Brief Title: Screening for Familial Colorectal Cancer (CRC) Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0316
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; CRC; Familial CRC; Cancer Screening; Questionnaire; First Degree Relatives; FDRs; Risk Communication
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Patients with Colorectal Cancer and their First Degree Relatives (FDRs).
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire regarding awareness of screening tests and attitudes toward colorectal cancer screening, taking 30-45 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this psychosocial research study is to learn about the knowledge, beliefs, and attitudes that people have toward screening for colorectal cancer. Another goal is to study how families communicate about colorectal cancer risk and colorectal cancer screening, with each other and with health care providers.

Objectives:

1. To evaluate psychosocial and external factors influencing colorectal cancer (CRC) patients' communication with their first-degree relatives (FDRs) about CRC risk and screening information.

   Using measures of knowledge, health beliefs and behavior, family closeness, openness and motivation to discuss CRC and screening, distress, provider support and background variables (sociodemographics, access to care, and medical history), we will conduct a cross-sectional study to evaluate factors influencing CRC patients' communication about CRC risk and screening information to their FDRs.
2. To evaluate psychosocial and external factors associated with CRC screening behavior among first-degree relatives of CRC patients.

Using measures of knowledge, health beliefs and behavior, family closeness and subjective norms, distress, provider interactions, benefits/barriers, and background variables (race/ethnicity, sociodemographics, access to care, and medical history), we will conduct a cross-sectional study of FDRs of CRC patients recruited under Aim 1 to evaluate factors associated with CRC screening behavior (specifically, colonoscopy adherence).

DETAILED DESCRIPTION:
You will be interviewed by a member of the study staff over the telephone. You will be asked about your awareness of screening tests for colorectal cancer, and your attitudes toward colorectal cancer screening. You also will also be asked about your family's past use of these screening tests, and how you discuss colorectal cancer risk and screening with your family and health care providers. Some demographic information also will be collected (such as your age or marital status). The questionnaire will take between 30 and 45 minutes to complete.

Your answers to the questions and your personal information will be kept strictly confidential. Your questionnaire answers will be identified with a code number, rather than a name, so that you cannot be identified.

This is an investigational study. Up to 325 colorectal cancer patients and their close relatives may take part in the study. All will be enrolled MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer (CRC) Patients: CRC patients will be eligible if they:

   * have a diagnosis of colorectal adenocarcinoma at or before age 60, and were diagnosed between 6 and 12 months prior to being contacted about this study (to allow adequate time for dissemination of CRC risk to family members, and to avoid interference with care surrounding the initial diagnosis);
   * have at least one living FDR age 40 years or older;
   * can read and speak English.
2. FDRs of CRC Patients: FDRs will be eligible if they

   * are age 40 years or older;
   * can read and speak English.

Exclusion Criteria:

1. CRC Patients: CRC patients will be excluded if they:

   * have a history of a known hereditary CRC syndrome (e.g., HNPCC, familial polyposis) or inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease); or
   * have an ECOG PS>1.
2. FDRs of CRC patients: FDRs will be excluded if they:

   * have a history of a known hereditary CRC syndrome (e.g., HNPCC, familial polyposis) or inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease); or
   * have a personal history of colon polyps or of cancer diagnosed within 5 years prior to entry into the study, with the exception of nonmelanoma skin cancer.

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with diagnosis of Colorectal Cancer at or before age 60 years, and their First Degree Relatives (FDRs) who are age 40 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2008-01-29 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Psychosocial + External factors influencing CRC patients' communication with FDRs about CRC risk & screening information | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, MPH,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org